CLINICAL TRIAL: NCT02092844
Title: Cognitive Behavioral Therapy for Insomnia and Nocturnal Hot Flashes in Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-102; 1K23NR014008 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-03-20 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2016-10

CONDITIONS: Menopause; Insomnia; Hot Flashes
Keywords: Menopause; Insomnia; Hot Flashes
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for Menopausal Insomnia (CBTMI) (Experimental): CBTMI is a combination of Cognitive Behavioral Therapy for Insomnia (CBTI) and Cognitive Behavioral Therapy for Hot Flashes (CBTH).
  Interventions: Behavioral: CBT for Menopausal Insomnia (CBTMI)
- Enhanced Treatment as Usual (Placebo Comparator): In the Enhanced Treatment as Usual/Information Control group, participants continue with clinical care of their choosing, but will be enhanced by the provision of 3 American Academy of Sleep Medicine (AASM) brochures.
  Interventions: Behavioral: CBT for Menopausal Insomnia (CBTMI)

INTERVENTIONS:
Behavioral: CBT for Menopausal Insomnia (CBTMI) — Cognitive Behavioral Therapy for Menopausal Insomnia (CBTMI) includes education about sleep, sleep restriction, stimulus control, cognitive restructuring of sleep interfering thoughts, and relapse prevention; while also addressing women's beliefs about and reactions to hot flashes.

SUMMARY:
The primary aim of the current study is to evaluate the effectiveness of a Cognitive Behavioral Therapy intervention in the treatment of menopause-associated insomnia and nocturnal hot flashes.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a primary care-based intervention for insomnia and nocturnal hot flashes (nHF) in peri- and postmenopausal women. Menopause-associated insomnia is associated with adverse consequences including reduced quality of life, increased health care utilization, and risk for psychiatric disorders and medical conditions. The poor benefit/risk ratio of estrogen and progesterone replacement therapy and concerns about long-term effects of sedative hypnotics has left women desperate for new approaches to resolve menopause-related health problems, including poor sleep. The proposed intervention aims to develop and evaluate a much-needed safe treatment of menopause-associated insomnia that combines and enhances cognitive behavioral therapies for insomnia and hot flashes. To maximize the public health impact, improve access, and reduce treatment barriers (stigma and transportation issues), we propose to evaluate the efficacy and effectiveness of the intervention delivered by nurses in gynecology clinics, where women receive routine care. Primary outcomes, for which the study is optimally designed and sufficiently powered, are subjectively- and objectively-measured sleep and nHF.

The Aims of this research are to:

1. To explore feasibility, acceptability (willingness to be randomized and dropout rates) of CBTMI, and indications of efficacy/effectiveness of CBTMI in a randomized, placebo-controlled, pilot study.
2. To explore the effects of CBTMI on the number and duration of arousals/awakenings that follow nHFs. If effective, the intervention has the potential to improve the quality of life in peri- and postmenopausal women and reduce the significant costs to society.

ELIGIBILITY:
Inclusion Criteria:

* Women in menopausal transition (defined by standardized criteria as variable cycle length seven days different from their normal cycle or >2 skipped cycles and an interval of amenorrhea of 2-12 months) or postmenopausal (defined as >12 months since last menstrual period).
* Meet Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria for insomnia assessed by Duke Structured Interview for Sleep Disorders.
* Score >14 on the Insomnia Severity Index (ISI) or >8 on the Pittsburgh Sleep Quality Index (PSQI).
* Have at least one nocturnal hot flash/night sweat on 3 or more nights a week (based on 2 weeks of daily hot flash diaries).

Exclusion Criteria:

* Chemotherapy/radiation-induced menopause.
* Presence of any unstable medical disorder assessed by medical tracking form.
* Traumatic brain injury or cognitive impairment defined by a score < 25 on Mini Mental Status Exam.
* Evidence of recent severe mental health disorders (e.g., suicide attempt or psychiatric hospitalization in past 3 years).
* Presence of psychotic disorder, substance abuse or dependence, or bipolar disorder, assessed by MINI International Neuropsychiatric Inventory (to increase generalizability other psychiatric comorbidities will not be excluded).
* Recent initiation/change in existing treatments that may impact sleep or nocturnal hot flashes (recency is defined by: < 4 weeks for antidepressant, < 16 weeks for any psychotherapy, and <8 weeks for estrogen, progestin, or androgen).
* As needed use of hypnotic, over-the-counter, or herbal supplements known to affect sleep or hot flashes.
* The following comorbid sleep disorders based on structured diagnostic interview: narcolepsy, circadian rhythm disorder, restless less syndrome, periodic leg movement disorder (PLMD), obstructive sleep apnea (OSA), or positive screening PLMD (PLMI > 15) or OSA (AHI > 15) on polysomnography (PSG) following screening visit.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | ≤2 weeks after therapy completion
Hot Flash Severity Diaries | Baseline, Post treatment (≤2 weeks after therapy completion), 1 month and 3 month follow-up

SECONDARY OUTCOMES:
Menopause Quality of Life Scale total score | Baseline, Post-treatment (≤2 weeks after therapy completion), 1 month and 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sara Nowakowski, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States